CLINICAL TRIAL: NCT03265002
Title: Effects of Fibre on Intestinal Volume and Gas in Irritable Bowel Syndrome
Brief Title: Fibre and Gas in Irritable Bowel Syndrome
Acronym: EFIGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17056
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: fibre; inulin; psyllium; small bowel MRI
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Inulin; Psyllium

STUDY DESIGN:
Intervention Model Description: single-centre, 4 period, 4 treatment, placebo-controlled crossover trial.
Who Masked: Participant, Investigator
Masking Description: Participants will be blind to the fibre product taken on each study visit. Masking will be assisted by adding lemon juice to the vehicle drink.
  The staff responsible for preparing this food will be members of the digestive diseases unit at the NIHR Nottingham Biomedical Research Centre and will not be involved in the study otherwise. The investigators responsible for MRI and symptom analysis will be kept blind to the intervention as data will be coded by date of study day, rather than by product received. Additionally MRI data will be assigned a 'scanning number' through the Sir Peter Mansfield Imaging Centre. This will pseudo-anonymise MRI data within the study so that associations between participants and scans will not be immediately obvious.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Ingestion of 500ml water with 50ml lemon juice and 20g dextrose
  Interventions: Dietary Supplement: Placebo
- Inulin (Experimental): Ingestion of 500ml water with 50ml lemon juice and 20g inulin
  Interventions: Dietary Supplement: Inulin
- Psyllium (Active Comparator): Ingestion of 500ml water with 50ml lemon juice and 20g psyllium
  Interventions: Dietary Supplement: Psyllium
- Inulin and Psyllium (Active Comparator): Ingestion of 500ml water with 50ml lemon juice and 20g inulin and 20g psyllium
  Interventions: Dietary Supplement: Inulin and psyllium

INTERVENTIONS:
Dietary Supplement: Placebo — Ingestion of 500ml water with 50ml lemon juice and 20g dextrose
  Arms: Placebo
Dietary Supplement: Inulin — Ingestion of 500ml water with 50ml lemon juice and 20g inulin
  Arms: Inulin
Dietary Supplement: Psyllium — Ingestion of 500ml water with 50ml lemon juice and 20g psyllium
  Arms: Psyllium
Dietary Supplement: Inulin and psyllium — Ingestion of 500ml water with 50ml lemon juice and 20g inulin and 20g psyllium
  Arms: Inulin and Psyllium

SUMMARY:
The aim of the study is to investigate how dietary fibre combinations affects gut physiology, particularly colonic gas production. Comparisons will be made between a single fermentable fibre (inulin), a non-fermentable fibre (psyllium) and a combination of the two. The study will also explore differences in response between diarrhoea-predominant and constipation-predominant IBS (IBS-D and IBS-C) respectively.

The participants will have a preliminary meeting to ensure they are eligible, then will attend the MRI department on 4 occasions separated by at least 1 week. They will ingest a drink with the fibre product mixed in, and will have 8 MRI scans (each lasting approximately 15 minutes).

DETAILED DESCRIPTION:
The aim of the study is to investigate how dietary fibre combinations affects gut physiology, particularly colonic gas production. Comparisons will be made between a single fermentable fibre (inulin), a non-fermentable fibre (psyllium) and a combination of the two. The study will also explore differences in response between diarrhoea-predominant and constipation-predominant IBS (IBS-D and IBS-C) respectively.

This is a single-centre, 4-period, 4-treatment, placebo-controlled, crossover trial. Each treatment will be taken once by each participant, with randomisation of treatment order.

The staff responsible for preparing this food will be members of the digestive diseases unit at the NIHR Nottingham Biomedical Research Centre and will not be involved in the study otherwise. The investigators responsible for MRI and symptom analysis will be kept blind to the intervention as data will be coded by date of study day, rather than by product received. Additionally MRI data will be assigned a 'scanning number' through the Sir Peter Mansfield Imaging Centre. This will pseudo-anonymise MRI data within the study so that associations between participants and scans will not be immediately obvious.

Randomisation All participants will take all 4 fibre/ placebo preparations in this crossover trial but the order in which the participants take them will be randomised. The randomisation will be undertaken by a member of the research division who is independent of the study using the remote, online, open source software www.randomization.com. The resulting code will be retained by staff responsible for food preparation in paper form, and will not be shared with the investigator team. A paper copy will be kept by the CI in a sealed envelope.

On enrolment to the study, participants will be allotted the next available randomization sequence. No stratification is needed as in a crossover design participants act as their own controls. There will be a washout period of at least one week between each study day to minimise any carryover effect.

Expected duration of participant participation Study participants will be participating in the study for 6-8 weeks. Women will not be scanned during their menstrual period to avoid confounding of symptom responses.

The study consists of 5 visits to the Queens Medical Centre, Nottingham (QMC). Visits will be in University departments embedded in the hospital, either in the Nottingham Digestive Diseases Centre (NDDC) or the Level A annex of the Sir Peter Mansfield Imaging Centre (SPMIC).

The first visit will be to take consent, assess eligibility and record baseline covariates of interest. All subsequent visits will MRI study days, where participants will undergo a series of MRI scans and other assessments.

Visit 1 This visit will last around 30 minutes. The researcher will confirm that the potential participant has understood the information sheet and answer any remaining questions. The participant will then be assessed for eligibility against the criteria previously set out. If eligibility is confirmed, participants will be asked for details of current medication use including contraception, smoking status, and significant past medical history. Height and weight will be recorded. Participants will complete the Hospital Anxiety and Depression Scale and the Patient Health Questionnaire-12. These questionnaires measure psychological traits that have been associated with symptom response in IBS and so will be relevant covariates.

Participants will then begin a 7-day screening diary of bowel habit and symptoms. This will be used to confirm frequency of IBS symptoms and IBS subtype. Participants will complete the Rome IV diagnostic questionnaire as part of their eligibility assessment. If there is a discrepancy between diary data and participant report on the Rome IV questionnaire, then the PI may decide to exclude the participant. To reduce patient burden, it will be acceptable to return completed diaries by post (prepaid envelope), by electronic communication (scan or photo), or in person.

Participants will also be informed that their GP will be contacted, both to inform them of the subject's participation and to confirm medical details where required.

Once eligibility has been confirmed, the Participant will be enrolled and randomised to a sequence of treatments. These will be administered during Visits 2 - 5. Participants will be asked to minimise their intake of fermentable carbohydrates on the day preceding each of these visits in addition to having a standardised evening meal. A dietary advice sheet will be provided.

Visits 2 - 5: MRI Study Days MRI study days will take place in the level A annex of the SPMIC, in the QMC. Visits will be at least 1 week apart to minimise any carryover effect. Participants will fast from 8pm on the evening before the Study Day. Water will be permitted after 8pm. On the morning of the Study Day participants will not eat or drink, other than a few sips of water to assist swallowing of essential medicines.

It will be confirmed that participants remain safe, eligible and willing to take part. The participants will change into surgical scrubs, in line with scanning policy and will then complete the first set of assessments.

The assessments will be:

1. Report of gastrointestinal symptoms. Symptoms of wind/ flatulence, bloating and abdominal pain will be scored on a 7-point scale, 0 - 3 in half-integer intervals(5).
2. Measurement of breath hydrogen and methane content from a single forced exhalation, using the GastroCheck device (Bedfont, UK).
3. An MRI scan including various scan sequences (See MRI Analysis section)

After fasting assessment participants will ingest a Test Drink. This will comprise still water made up to 500mL with 50mL lemon juice (PLj, Holland&Barrett, UK), into which the test supplement will be mixed.

The Test Fibres used will be:

A. 20g Inulin B. 20g Inulin and 20g psyllium C. 20g psyllium D. 20g dextrose (0g fibre content - placebo control)

The test drink will be administered in 2 x 250mL portions to prevent swelling of fibres. Participants will be given 10 minutes to consume the total 500mls.

Assessments will be repeated immediately after ingestion, then at intervals post-ingestion as shown in the schematic. Breath symptoms will be measured every 30 minutes for 2 hours, then hourly. MRIs will be taken immediately post ingestion, then hourly for 6 hours. After 3 hours a meal will be provided, designed to be low in fermentable carbohydrate and fibre. This will stimulate gut motility and movement of small bowel content into the colon. The whole Study Day will last around 8 hours.

At the end of the Study Day participants will be asked for an overall rating of their symptoms throughout the day, and an assessment of product acceptability on the basis of their experience (0 - 100 visual analogue scale).

In between assessments participants will be provided with a comfortable sitting area which is part of the level A annex. The participants will be advised to bring material such as magazines, books or electronic devices for entertainment. Guest access to the university's wireless internet (wifi) network will be available.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Fulfilment of the Rome IV criteria for Irritable Bowel Syndrome for at least 3 months:

  * Abdominal pain at least two or more days per week.
  * Pain associated with two or more of the following:

    * Related to defecation on at least ≥30% of occasions
    * Associated with a change in frequency of stool on ≥30% of occasions
    * Associated with a change in form (appearance) of stool on ≥30% of occasions
  * Symptom onset at least 6 months prior to diagnosis

Exclusion Criteria:

* Pregnancy declared by candidate
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Inability to lie flat or exceed scanner limits of weight <120kg
* Unwilling to cease use of supplementary fibre or osmotic laxatives for the duration of the study
* Unable to stop drugs known to alter GI motility or transit including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists or osmotic laxatives for 2 days before, and during, MRI study days.

  * Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria
* Reported alcohol intake of >28 units/ week with daily drinking
* Intention to change smoking behaviour during the study
* History declared by the candidate of other pre-existing gastrointestinal disorders, including but not limited to:

  * Inflammatory Bowel Disease
  * Coeliac Disease
  * Pancreatitis
  * Gallstone disease (biliary colic, cholecystitis; asymptomatic presence of gallstones permitted)
  * Complicated diverticulitis (asymptomatic presence of diverticula permitted)
  * Cancer of the gastrointestinal tract
  * Gastroparesis
  * Other functional gastrointestinal disorders will be permitted as they frequently co-exist with IBS.
* Any reported history of gastrointestinal resection (excluding appendicectomy or cholecystectomy)
* Presence of an intestinal stoma
* Poor understanding of English language
* Participation of any medical trials for the past 3 months
* Judgement by the PI that the candidate who will be unable to comply with the full study protocol e.g. Diabetes, severe COPD

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in colonic gas | baseline, 0, 1, 2, 3, 4, 5 and 6 hours post ingestion of the fibre drink
  in arbitrary units measured by MRI

SECONDARY OUTCOMES:
Change from the baseline in colonic volume | baseline, 0, 1, 2, 3, 4, 5 and 6 hours post ingestion of the fibre drink
  in mL measured by MRI
Change from the baseline in small bowel water content | baseline, 0, 1, 2, 3, 4, 5 and 6 hours post ingestion of the fibre drink
  in mL measured by MRI
Change from the baseline in breath hydrogen | baseline, 0mins, 30mins, 1 hour, 90mins, 2 hours, 3, 4, 5 and 6 hours post ingestion of fibre drink
  in parts per million using the GastroCheck device
Change from the baseline in severity of pain, bloating and flatulence | baseline, 0mins, 30mins, 1 hour, 90mins, 2 hours, 3, 4, 5 and 6 hours post ingestion of fibre drink
  assessed by the Gastrointestinal Symptom Rating Scale, using a 7-point scale

OTHER OUTCOMES:
Product acceptability | throughout the study completion, measured after the 6 hour postprandial measurements.
  gained by questionnaire
Change from the baseline in contractility of the ascending colon | baseline, 0, 1, 2, 3, 4, 5 and 6 hours post ingestion of the fibre drink
  assessed by the MRI motility index
breath methane | baseline, 0mins, 30mins, 1 hour, 90mins, 2 hours, 3, 4, 5 and 6 hours post ingestion of fibre drink
  in parts per million using the GastroCheck device

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, Ph, BMBS, Study Chair — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Major G, Pritchard S, Murray K, Alappadan JP, Hoad CL, Marciani L, Gowland P, Spiller R. Colon Hypersensitivity to Distension, Rather Than Excessive Gas Production, Produces Carbohydrate-Related Symptoms in Individuals With Irritable Bowel Syndrome. Gastroenterology. 2017 Jan;152(1):124-133.e2. doi: 10.1053/j.gastro.2016.09.062. Epub 2016 Oct 14. PMID 27746233
- [Derived] Gunn D, Abbas Z, Harris HC, Major G, Hoad C, Gowland P, Marciani L, Gill SK, Warren FJ, Rossi M, Remes-Troche JM, Whelan K, Spiller RC. Psyllium reduces inulin-induced colonic gas production in IBS: MRI and in vitro fermentation studies. Gut. 2022 May;71(5):919-927. doi: 10.1136/gutjnl-2021-324784. Epub 2021 Aug 5. PMID 34353864